CLINICAL TRIAL: NCT00120003
Title: Scandinavian Candesartan Acute Stroke Trial
Brief Title: Scandinavian Candesartan Acute Stroke Trial (SCAST)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ullevaal University Hospital (Other)
Collaborators: Southern-Eastern Norway Health Authorities RHF (Unknown); AstraZeneca (Industry); Takeda (Industry)
Responsible Party: Director of Research Andreas Moan, Ullevaal University Hospital
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 050321
Record Dates: First submitted 2005-07-06; First posted 2005-07-14 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2006-09

CONDITIONS: Stroke
Keywords: Acute stroke; Elevated blood pressure; Blood pressure lowering treatment
MeSH Terms: conditions — Stroke; Hypertension | interventions — candesartan cilexetil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Candesartan Cilexetil (Experimental): Candesartan Cilexetil
  Interventions: Drug: Candesartan Cilexetil
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Candesartan Cilexetil — 4 mg on day 1; 8 mg on day 2; 16 mg on days 3-7
  Arms: Candesartan Cilexetil
Drug: Placebo — 4 mg on day 1; 8 mg on day 2; 16 mg on days 3-7
  Arms: Placebo

SUMMARY:
The purpose of this trial is to assess whether the blood pressure lowering agent candesartan (an angiotensin receptor type 1 blocker) is effective when given to patients with acute stroke and elevated blood pressure.

Hypothesis:

AT1 receptor blockade with candesartan in acute stroke will:

1. reduce the risk of death or major disability at 6 months by a 6% absolute risk reduction, relative to placebo.
2. reduce the risk of the combined event of "vascular" death, myocardial infarction, or stroke during the first 6 months by a 25% relative risk reduction, relative to placebo

DETAILED DESCRIPTION:
It has long been a controversy whether elevated blood pressure should be lowered in the acute phase of stroke. Current clinical practice is generally to accept high blood pressure in the acute phase of stroke, to avoid reduction of cerebral blood perfusion. This practice has a well-founded theoretical basis, but is not supported by evidence from clinical trials. The newly published study ACCESS (Stroke 2003;34:1699) showed a clear beneficial effect of the angiotensin receptor blocker candesartan in the acute phase of stroke, but the trial was seriously underpowered.

The Scandinavian Candesartan Acute Stroke Trial (SCAST) is designed to provide reliable data on the effects of candesartan in a wide variety of patients with acute stroke (target recruitment 2,500). Patients presenting with acute stroke (<30 hours) and systolic blood pressure ≥140 mm Hg will be randomly assigned to candesartan 4 to 16 mg once daily or matching placebo for 7 days, followed by candesartan treatment for 6 months for patients who are hypertensive at the end of the treatment period (at clinician's discretion). Follow-up will be performed double-blind at 30 days, 3 months and 6 months.

The trial is co-ordinated from Ullevaal University Hospital in Oslo, Norway. Over 100 centres from Norway, Sweden, Denmark and Belgium have agreed to participate. Financial contributors: The Eastern Norway Regional Health Authority, AstraZeneca, and Ullevaal University Hospital (Oslo). AstraZeneca will supply drugs and placebo for the trial.

ELIGIBILITY:
Inclusion Criteria:

* Clinical stroke syndrome with limb paresis, not likely to represent a transient ischaemic attack or non-stroke pathology (e.g. cerebral tumour)
* Systolic blood pressure ≥ 140 mm Hg
* Trial treatment possible within 30 hrs of symptom onset. If time of onset is not known, use the time when the patient was last known to be well.
* Consent (subsidiary, assent from legal acceptable representative, or waiver of consent)
* Age >18 years

Exclusion Criteria:

* Markedly reduced consciousness (i.e. Scandinavian Stroke Scale consciousness score ≤ 2)
* Patient already receiving AT1 receptor blocker
* Contraindication to treatment with AT1 receptor blocker, e.g.:

  * known renal failure (women: creatinine ≥ 150 µmol/L; men: ≥ 180 µmol/L)
  * previously diagnosed bilateral renal artery stenosis
  * previously diagnosed high-grade aortic stenosis
  * previously diagnosed seriously impaired liver function and/or cholestasis
  * known intolerance to candesartan or other tablet ingredients
* Clear indication, in the clinician's view, for start of treatment with AT1 receptor blocker during the treatment period (e.g. chronic heart failure grade III-IV, in the presence of intolerance to ACE inhibitors)
* Clear indication, in the clinician's view, for antihypertensive therapy during the acute phase of stroke (i.e. concurrent hypertensive encephalopathy or aortic dissection, or other situations)
* Other serious or life-threatening disease before the stroke:
* Patient severely mentally or physically disabled (e.g. Mini Mental Status score < 20, or modified Rankin Scale score ≥ 4)
* Life expectancy < 12 months
* Patient unavailable for follow-up (e.g. no fixed address)
* Pregnant or breast-feeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2005-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Death or major disability (defined by the modified Rankin scale) at 6 months | 6 months
The composite event "vascular" death, myocardial infarction, or stroke during the first 6 months | 6 months

SECONDARY OUTCOMES:
Scandinavian Stroke Scale score at 7 days | 7 days
Barthel Index score at 6 months | 6 months
EuroQol score at 6 months | 6 months
Mini-Mental State score at 6 months | 6 months
Death (all-cause death and "vascular" death) | 6 months
Recurrent stroke (ischaemic, haemorrhagic, or unspecified) | 6 months
Myocardial infarction | 6 months
Combination of the above events | 6 months
Symptomatic hypotension | 7 days
Renal failure | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Eivind Berge, MD, PhD, Principal Investigator — Ullevaal University Hospital; Per Morten Sandset, Prof, Study Chair — Ullevaal University Hospital; Povel Paus, MD, PhD, Study Director — Ullevaal University Hospital
Locations (1):
- Ullevaal University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Wang X, Moullaali TJ, Li Q, Berge E, Robinson TG, Lindley R, Zheng D, Delcourt C, Arima H, Song L, Chen X, Yang J, Chalmers J, Anderson CS, Sandset EC. Utility-Weighted Modified Rankin Scale Scores for the Assessment of Stroke Outcome: Pooled Analysis of 20 000+ Patients. Stroke. 2020 Aug;51(8):2411-2417. doi: 10.1161/STROKEAHA.119.028523. Epub 2020 Jul 9. PMID 32640944
- [Derived] Berge E, Cohen G, Lindley RI, Sandercock P, Wardlaw JM, Sandset EC, Whiteley W. Effects of Blood Pressure and Blood Pressure-Lowering Treatment During the First 24 Hours Among Patients in the Third International Stroke Trial of Thrombolytic Treatment for Acute Ischemic Stroke. Stroke. 2015 Dec;46(12):3362-9. doi: 10.1161/STROKEAHA.115.010319. Epub 2015 Oct 20. PMID 26486868
- [Derived] Hornslien AG, Sandset EC, Igland J, Terent A, Boysen G, Bath PM, Murray GD, Berge E. Effects of candesartan in acute stroke on vascular events during long-term follow-up: results from the Scandinavian Candesartan Acute Stroke Trial (SCAST). Int J Stroke. 2015 Aug;10(6):830-5. doi: 10.1111/ijs.12477. Epub 2015 Mar 22. PMID 25808741
- [Derived] Sandset EC, Jusufovic M, Sandset PM, Bath PM, Berge E; SCAST Study Group. Effects of blood pressure-lowering treatment in different subtypes of acute ischemic stroke. Stroke. 2015 Mar;46(3):877-9. doi: 10.1161/STROKEAHA.114.008512. Epub 2015 Feb 5. PMID 25657183
- [Derived] Jusufovic M, Sandset EC, Bath PM, Berge E; Scandinavian Candesartan Acute Stroke Trial Study Group. Blood pressure-lowering treatment with candesartan in patients with acute hemorrhagic stroke. Stroke. 2014 Nov;45(11):3440-2. doi: 10.1161/STROKEAHA.114.006433. Epub 2014 Sep 25. PMID 25256183
- [Derived] Hornslien AG, Sandset EC, Bath PM, Wyller TB, Berge E; Scandinavian Candesartan Acute Stroke Trial Study Group. Effects of candesartan in acute stroke on cognitive function and quality of life: results from the Scandinavian Candesartan Acute Stroke Trial. Stroke. 2013 Jul;44(7):2022-4. doi: 10.1161/STROKEAHA.113.001022. Epub 2013 May 9. PMID 23660849
- [Derived] Sandset EC, Murray GD, Bath PM, Kjeldsen SE, Berge E; Scandinavian Candesartan Acute Stroke Trial (SCAST) Study Group. Relation between change in blood pressure in acute stroke and risk of early adverse events and poor outcome. Stroke. 2012 Aug;43(8):2108-14. doi: 10.1161/STROKEAHA.111.647362. Epub 2012 May 24. PMID 22627991
- [Derived] Sandset EC, Bath PM, Boysen G, Jatuzis D, Korv J, Luders S, Murray GD, Richter PS, Roine RO, Terent A, Thijs V, Berge E; SCAST Study Group. The angiotensin-receptor blocker candesartan for treatment of acute stroke (SCAST): a randomised, placebo-controlled, double-blind trial. Lancet. 2011 Feb 26;377(9767):741-50. doi: 10.1016/S0140-6736(11)60104-9. PMID 21316752
- [Derived] Sandset EC, Murray G, Boysen G, Jatuzis D, Korv J, Luders S, Richter PS, Roine RO, Terent A, Thijs V, Berge E; SCAST Study Group. Angiotensin receptor blockade in acute stroke. The Scandinavian Candesartan Acute Stroke Trial: rationale, methods and design of a multicentre, randomised- and placebo-controlled clinical trial (NCT00120003). Int J Stroke. 2010 Oct;5(5):423-7. doi: 10.1111/j.1747-4949.2010.00473.x. PMID 20854630
- See also: Click here for more information about this trial — http://www.scast.no